CLINICAL TRIAL: NCT07054827
Title: Effect of Intradialytic Resistance Versus Aerobic Exercise on Cardiovascular System in Patients on Regular Hemodialysis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Mahmoud Gouda, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005770
Record Dates: First submitted 2025-06-28; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Hemodialysis Complication
MeSH Terms: interventions — Renal Dialysis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medical therapy group (Active Comparator): Patients with chronic kidney disease will receive hemodialysis only, for four hours, 3 times per week.
  Interventions: Other: Hemodialysis
- intra-dialytic resistive exercise group (Experimental): Patients with chronic kidney disease will receive an intra-dialytic resistance exercise for 12 weeks (3 sessions/week) in addition to hemodialysis.
  Interventions: Other: Hemodialysis; Other: Intradialytic resistive exercise
- intra-dialytic aerobic exercise group (Experimental): Patients with chronic kidney disease will receive an intra-dialytic aerobic exercise (leg pedaling) for 12 weeks (3 sessions/week) in addition to hemodialysis.
  Interventions: Other: Hemodialysis; Other: Intradialytic aerobic exercise

INTERVENTIONS:
Other: Hemodialysis — The participants receive hemodialysis for 4 hours, 3 times per week
Other: Intradialytic resistive exercise — The participants will receive intradialytic resistive exercise for 12 weeks (3 sessions/ week).
  Duration: 30 minutes during the first 2 hours of each dialysis session in a recumbent position or seated position.
  Time of session: The program starts with a warm-up phase which is 3:5 minutes in the form of light aerobic and stretching exercises for big muscles and ends with a cooling down phase which is 3:5 in the form of light aerobic exercise.
  The resistance exercises include exercises for the big muscles of only the Lower Limbs (LL) muscles of single and multiple-joint which are:1- Knee extensors, 2- Knee flexors, 3- Hip flexors, 4- Hip abductors and adductors. using sandbags of different weights. Sandbag weights are placed on the distal third of the tibia for LL exercises.
  Intensity: On the Borg's Scale of Perceived Exertion, which will be measured every 5 minutes during exercise.
  Arms: intra-dialytic resistive exercise group
Other: Intradialytic aerobic exercise — Patients with chronic kidney disease will receive an intradialytic aerobic exercise for 12 weeks (3 sessions/ week).
  Duration: 30 minutes during the first 2 hours of each dialysis session using a stationary bicycle ergometer in a supine position or seated position.
  Time of session: The warming up and the cooling down phase consists of 5:10 minutes of slow Pedaling. the main exercise phase consisted of 20 minutes of cycling.
  Intensity: The use of the Borg's Scale of Perceived Exertion (RPE) scale enables the intensity of the exercise to be adapted According to the tolerance of each patient.
  The use of the RPE scale enables the intensity of the exercise to be adapted According to the tolerance of each patient, the aim was to obtain between 11 light And 14 somewhat hard.
  Arms: intra-dialytic aerobic exercise group

SUMMARY:
The purpose of the study is to compare the effect of resistance exercise and aerobic exercise on intradialytic hypotension in patients undergoing hemodialysis.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is one of the leading causes of global morbidity and mortality. In the 2019 Global Burden of Disease study, CKD was among the top ten risks associated with the highest number of deaths worldwide, with a death toll of 3.16 million deaths.

Patients undergoing dialysis in Egypt in 2020 are mostly men (59%), and half of them are aged ≥55 years. Hypertension is the most common cause of end-stage kidney disease at 41%, followed by diabetes at 14%, whereas glomerulonephritis is the primary diagnosis in 3% of patients undergoing dialysis.

Hemodialysis (HD), continuous ambulatory peritoneal dialysis, and kidney transplantation are the three main modalities of renal replacement therapy. Hypotension is the most reported complication of routine outpatient HD treatments.

Toxic substances, also called uremic toxins, in the blood result in malaise, paraesthesia, mental impairment, peripheral circulatory disturbance, and muscle dysfunction.

While patients exercise during dialysis, those toxins move through the dialyzer with a large flux from the tissue to the vascular compartment. It results in increased muscle blood flow and opened capillary surface area. Besides, the intradialytic exercise showed not only better adoption and adherence but also a lower drop-out and greater compliance.

So, this study will investigate the effect of resistance and aerobic exercises on intradialytic hypotension in patients undergoing hemodialysis. thus, may affect the quality of life in chronic kidney disease dialysis patients. The results of this study may shed light on which of the selected exercises can decrease the risk of Intradialytic hypotension to help dialysis patients. To our knowledge, there are no previous similar studies.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease (ESRD) or stage 5 chronic kidney disease (CKD) in which on maintenance regular HD (three sessions/week (on alternate days), for four hours/session for more than a year to five years when starting the study.
* Both gender male and female aged from 45 to 60 years old.
* Patients with intradialytic hypotension sudden drops of systolic pressure of more than 20 mm Hg or diastolic pressure of more than 10 mmHg.
* Receiving hemodialysis (HD) through uncomplicated arm arteriovenous (A-V) fistula.
* Patients with Body Mass Index (BMI): 18,5 < 30kg/m2.
* In a stable medical, clinical, and hemodynamic condition
* Untrained at baseline and did not participate in any regular physical activity before.

Exclusion Criteria:

* Severe Chest diseases (either obstructive or restrictive).
* Clinical signs of a severe cardiac event. (eg, severe atherosclerosis, congestive heart failure),
* Severe psychiatric or cognitive impairment, who unable to follow comment.
* Neurological disorders affecting respiratory muscles or any muscular dystrophies (cervical disc or bulge).
* Patients with severe self-limiting illness (e.g., cancer).
* Patients with Body Mass Index (BMI) > 30kg/m2.
* Previous renal transplantation patients.
* Pregnant females or became pregnant during the study.
* Patients started HD in less than a year or more than 5 years.
* Hospitalized during the prior month.
* Patients who were irregular in HD or not adherent to the exercise program.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-07-05 (Estimated); Primary Completion 2025-11-05 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure measurement | 12 weeks
  Blood pressure (BP) will be measured on the non-access arm using automatic BP cuffs attached to the patient's hemodialysis machine which is used routinely at each respective hemodialysis clinic. As well as for ankle brachial pressure index. Systolic blood pressure measurements will be taken pre-hemodialysis, at hemodialysis start (baseline), post-hemodialysis, and every 15 minutes during each dialysis session. BP measurements will be taken before selected exercise and after exercise.
Diastolic blood pressure measurement | 12 weeks
  Blood pressure (BP) will be measured on the non-access arm using automatic BP cuffs attached to the patient's hemodialysis machine which is used routinely at each respective hemodialysis clinic. As well as for ankle brachial pressure index. diastolic blood pressure measurements will be taken pre-hemodialysis, at hemodialysis start (baseline), post-hemodialysis, and every 15 minutes during each dialysis session. BP measurements will be taken before selected exercise and after exercise.
Ankle-Brachial Index (ABI) | 12 weeks
  This non-invasive test compares blood pressure in the ankles to blood pressure in the arms. An ABI below 0.9 usually suggests peripheral artery disease (PAD), a common cause of circulatory issues.
Peripheral oxygen saturation | 12 weeks
  Pulse oximetry is a non-invasive method used to measure the oxygen saturation level (SpO2) in the blood, providing an estimate of how much oxygen the hemoglobin in red blood cells is carrying. It provides data on oxygen delivery to extremities, which may be impaired in circulation issues. Normally, its value is 95-99%.
Creatinine level | 12 weeks
  Blood analysis will be used to measure creatinine level for all patients before and after intervention. Its values vary by sex; 0.6-1.2 mg/dl for men and 0.5-1.1 mg/dl for women.
blood urea level | 12 weeks
  Blood analysis will be used to measure blood urea for all patients before and after intervention. its normal value ranges from 17-43 mg/dl.
blood urea nitrogen test | 12 weeks
  Blood analysis will be used to measure blood urea nitrogen for all patients before and after intervention. its normal value ranges from 7-20 mg/dl.
serum albumin | 12 weeks
  Blood analysis will be used to measure serum albumin for all patients before and after intervention. its normal value in adults is typically 3.5-5.0 g/L.

SECONDARY OUTCOMES:
Six minutes walking Test (6 MWT) | 12 weeks
  A 6-minute walk test (6MWT) is a major physical test in the dialysis population. Its value lies in the fact that it is a self-paced test of walking capacity and functional ability of daily physical activities which are mostly performed at submaximal level of exertion.
  6MWT is a major physical tests in dialysis population. Its value lies in the fact that it is a self-paced test of walking capacity and reflects the functional ability at daily physical activities which are mostly performed at submaximal level of exertion. It is carried out in a 30 m long corridor. Subjects will be instructed to walk from end to end of the corridor and to cover the greatest distance possible in six minutes. Patients who need rest due to dyspnea will be instructed to continue walking as soon as they feel able, but the timer doesn't stop.
The Kidney Disease Quality of Life Short Form (KDQOL-SF) | 12 weeks
  is a self-reported measure of health that particularly concerns individuals with chronic kidney disease (CKD). The KDQOL-36 is a short version of KDQOL-SF that includes only 36 questions.
  The survey can be administered in 3-5 min, which saves both time and resources. Each subscale score ranges between 0 and 100, with increasing values equating to better health.

CONTACTS AND LOCATIONS:
Overall Officials: Sahier El-Khashab, Professor, Study Director — Cairo University; Nagwa Badr, Professor, Study Chair — Cairo University
Locations (1):
- Yasmin Mohamed Mahmoud Gouda, Cairo, Egypt